CLINICAL TRIAL: NCT00035841
Title: Phase 2 Study of TLK286 in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Telik (Industry)
Responsible Party: Gail Brown, M.D. Chief Medical Officer, Telik, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK286.2008
Record Dates: First submitted 2002-05-06; First posted 2002-05-07 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — TER 286

INTERVENTIONS:
Drug: TLK286

SUMMARY:
The purpose of this study is to determine the effectiveness of TLK286 in treatment of metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of breast cancer
* Metastatic disease
* Measurable or evaluable disease
* No prior chemotherapy regimens
* Age at least 18 years
* Adequate liver and kidney function
* Adequate bone marrow function

Exclusion Criteria:

* Pregnant or lactating women
* Unstable medical conditions
* Chemotherapy within 14 days of TLK286
* Radiation therapy within 14 days of TLK286
* Hormonal therapy within 14 days of TLK286
* Immunotherapy within 14 days of TLK286
* CNS metastasis unless controlled by treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-04; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Arizona Cancer Center, Tucson, Arizona
  - Indiana University Medical Center, Indianapolis, Indiana
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio